CLINICAL TRIAL: NCT03113708
Title: The Effect of Heparinization Due to LBW in Cardiac Surgery
Brief Title: The Effect of Heparinization Due to LBW
Acronym: LBWH
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Adiyaman University Research Hospital (Other)
Responsible Party: Principal Investigator, Dr. Ülkü Sabuncu, Medical Doctor, Adiyaman University Research Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: LBW heparin
Record Dates: First submitted 2017-03-25; First posted 2017-04-13 (Actual); Last update posted 2017-04-14 (Actual); Status verified 2017-04

CONDITIONS: Heparin; Heparin Overdose; Bleeding
Keywords: heparin; heparin antagonists; cardiac surgery; active clotting time
MeSH Terms: conditions — Hemorrhage | interventions — Heparin

STUDY DESIGN:
Who Masked: Care Provider
Masking Description: Closed envelope
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Heparinisation,actual body weight (Sham Comparator): In 'Heparinisation,actual body weight' group , heparin sodium; will be done according to actual body weight and ACT will be recorded prior to CPB. Before coming out CPB, protamine will be done according to heparin dose. And then ACT will be recorded.
  Interventions: Drug: Heparin Sodium
- Heparinisation, lean body weight (Experimental): In 'Heparinisation, lean body weight' group heparin sodium will be done according to lean body weight and ACT will be recorded prior to CPB. Before coming out CPB, protamine will be done according to heparin dose. And then ACT will be recorded.
  Interventions: Drug: Heparin Sodium

INTERVENTIONS:
Drug: Heparin Sodium — Heparinisation 2-4 mg/kg will be done according to actual body weight or lean body weight.

SUMMARY:
High dose heparin regimens are required in cardiac surgery under cardiopulmonary bypass (CPB) and this may increase postoperative bleeding. The aim of this study is to evaluate the effect of heparin dose calculated according to lean body weight on intraoperative and postoperative bleeding.

DETAILED DESCRIPTION:
Patients with preoperative demographic data such as age, gender, body weight, height, and additional disease, medications, previous surgery, preoperative Htc / Hb values were recorded in the operation room without medical premedication. Standard anesthesia induction was performed after arterial cannulation and peripheral venous route. Patients were randomly divided into two groups: 400 IU heparin / kg (Group I) and 400 IU heparin / kg (Group II) according to actual body weight and lean body weight respectively before CPB. Before and after heparin administration, CPB entry and ACT (Activated Clotting Time) values were counted every 30 minutes, after CPB exit and protamine. In both groups, supplemental heparin was administered when there was a failure to reach the pre-CPB target ACT value of 400 sec. Hemodynamic data and transfusion requirements were recorded during the operation. Patient's intraoperative CPB and crossover times, postoperative drainage volume and blood transfusion requirement were recorded.

ELIGIBILITY:
Inclusion Criteria:

* 18-65 years old, first time valve surgeries which was done on-pump.

Exclusion Criteria:

* Revision valve surgeries
* Patients with coagulation deficits

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2017-04-30 (Estimated); Primary Completion 2017-05-20 (Estimated); Study Completion 2017-06-20 (Estimated)

PRIMARY OUTCOMES:
ACT | Through study completion, an average of 48 hours
  Activated clotting time

SECONDARY OUTCOMES:
Bleeding | Through study completion, an average of 48 hours
  Postoperative bleeding

CONTACTS AND LOCATIONS:
Overall Officials: Ulku Sabuncu, Principal Investigator — Yuksek Ihtisas Hospital

IPD SHARING:
Plan to Share IPD: No